CLINICAL TRIAL: NCT05998707
Title: The Application of the New Magnetic Resonance Technique-UTE in Thoracic Lesions
Brief Title: The Application of the New Magnetic Resonance UTE Technique in Thoracic Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: ZDWY.FSK.024
Record Dates: First submitted 2023-08-02; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Lung Diseases
Keywords: Lung mass, UTE, ZTE, nodule, MRI
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- benign group: benign lesions in the lung
- malignant group: malignant tumor in the lung

SUMMARY:
Quantitative characteristic values of lung lesions were obtained by UTE technique, so as to make qualitative diagnosis of benign and malignant lesions. And to explore the clinical feasibility of CT-like technology - high resolution ZTE technology in the diagnosis of pulmonary diseases.

DETAILED DESCRIPTION:
Ultrashort echo time (UTE) sequence can obtain data from T2* for lung imaging before T2* decays in lung parenchyma with extremely short echo time, which makes up for the defect that conventional MRI cannot clearly display short T2 tissue imaging, and can provide more supplementary information for lung CT scan. There has been a lot of research progress in the evaluation of neonatal lung disease, chronic obstructive airway disease and pneumonia. The 3D UTE sequence developed on this basis has made great progress in improving the resolution, signal-to-noise ratio and shortening the scanning time of lung MR Images, and has successfully obtained submillimeter high-resolution images. The purpose of this study was to explore the value of MRI ultra-short echo technology in the qualitative diagnosis of benign and malignant lung lesions, and to explore the clinical application of CT-like technology - high resolution ZTE technology in the lung.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. There are lung lesions, and the solid component is ≥6mm;
3. Chest CT plain scan or /+ enhanced examination within 4 weeks.

Exclusion Criteria:

1. There are metal implants in the corresponding parts of the chest;
2. MRI contrast agent allergy;
3. Claustrophobia;
4. Pregnant women;
5. High fever;
6. Respiratory failure;
7. Lung lesion biopsy within 4 weeks prior to examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-13 (Estimated); Study Completion 2024-06-13 (Estimated)

PRIMARY OUTCOMES:
proton density fat fraction (PDFF) | baseline (before surgery)
  Determination of proton density fat fraction by magnetic resonance imaging
T2 relaxation rate | baseline (before surgery)
  R2*
Magnetization Transfer Ratio (MTR) | baseline (before surgery)
  Magnetization Transfer Ratio

SECONDARY OUTCOMES:
Subjective rating | baseline (before surgery)
  rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Shaolin Li, Study Director — Fifth Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Radiography department, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No